CLINICAL TRIAL: NCT00692562
Title: Simultaneous Islet-Kidney Transplantation in Patients of Type 1 Diabetes With End-stage Renal Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: FUZHOU GENERAL HOSPITAL, FUZHOU GENERAL HOSPITAL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIK2005
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2008-06

CONDITIONS: Type 1 Diabetes Mellitus; End-stage Renal Disease
Keywords: Islets of Langerhans Transplantation; Kidney Transplantation; Type 1 Diabetes Mellitus; alemtuzumab
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Procedure: simultaneous islet-kidney transplantation

INTERVENTIONS:
Procedure: simultaneous islet-kidney transplantation

SUMMARY:
The aim of this study was to evaluate the efficiency and safety of simultaneous islet-kidney transplantation in patients of type 1 diabetes with end-stage renal disease using a glucocorticoid-free immunosuppressive regimen with alemtuzumab induction. Islet transplantation can result in insulin independence with excellent metabolic control when glucocorticoid-free immunosuppression is combined with the infusion of an adequate islet mass. Alemtuzumab (Campath-1H ®) is a 150-kDa humanized IgG1 monoclonal antibody that targets the CD52 antigen. Prolonged lymphocyte depletion can be expected following alemtuzumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 to 60 years of age.
* Ability to provide written informed consent.
* Clinical history compatible with type 1 diabetes (T1DM) as defined by the WHO guidelines(1999) on the Diagnosis and classification of Diabetes Mellitus.
* manifest signs and symptoms that are severe enough to be incapacitating.
* Basal C-peptide<0.5ng/mL
* patients with poor diabetes control (HbA1c >7% but <12%)
* progressive diabetic complications.
* end-stage renal disease(serum creatinine>450μmol/l)

Exclusion Criteria:

* age <18 years or >60 years
* diabetic history <5 years
* BMI>27
* body weight >80kg
* exogenous insulin requirement >1 unit/kg/day
* severe anemia (male <8g/dl, female <7g/dl)
* low white blood cell count (<3000/dl)
* liver dysfunction
* Symptomatic peptic ulcer disease
* Any malignancy
* Active infection including hepatitis B, hepatitis C, HIV, or TB
* panel reactive antibody >20%
* Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2005-06; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Exogenous insulin requirement | 5
kidney function | 5

SECONDARY OUTCOMES:
Hemoglobin A1c | 5
Glucose and C-peptide levels | 5
Portal vein Ultrasound | 1
liver function | 5
Complete Blood Count | 5
autoantibodies | 5

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Tan, professor, Principal Investigator — Fuzhou General Hospital
Locations (1):
- Fuzhou General Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Tan J, Yang S, Cai J, Guo J, Huang L, Wu Z, Chen J, Liao L. Simultaneous islet and kidney transplantation in seven patients with type 1 diabetes and end-stage renal disease using a glucocorticoid-free immunosuppressive regimen with alemtuzumab induction. Diabetes. 2008 Oct;57(10):2666-71. doi: 10.2337/db08-0358. Epub 2008 Jul 15. PMID 18633105